CLINICAL TRIAL: NCT04863066
Title: A Phase I Trial Using Third-Generation CAR-T-cell Therapy in Individuals With HIV-1 Infection
Brief Title: Third-Generation CAR-T-cell Therapy in Individuals With HIV-1 Infection
Acronym: TCTIWHI
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing 302 Hospital (Other)
Collaborators: Tsinghua University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-HIV-001
Record Dates: First submitted 2020-12-07; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2020-10

CONDITIONS: HIV-1
Keywords: CAR T cells; HIV-1 infection; safety; HIV latent reservoir
MeSH Terms: interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-T-cell therapy (Experimental): Four patients with plasma HIV RNA <50 copies/ml and CD4+T cell count more than 350 cells/μl receiving at least one-year antiviral treatment are injected intravenously with 1×10^5 CAR-T cells/kg body weight. If the dosage of 1×10^5 CAR-T cells/kg body weight is well tolerated, 5×10^5 CAR-T cells/kg body weight will be infused for another 4 subjects who meet the inclusion and exclusion criteria.
  Interventions: Biological: CAR-T cells

INTERVENTIONS:
Biological: CAR-T cells — The presence of latent infected cells remains a key barrier to HIV-1 functional cure. Current approach to reducing the latent HIV reservoir is to reactivate virus-containing cells to make them be detected and eliminated by host defense. Endogenous cytotoxic T-lymphocytes (CTL) may not be adequate because of cellular exhaustion and immune escape of virus. We have designed a kind of CAR-T cell based on CTL engineered to express a scFv of a broadly neutralizing anti-HIV antibody. According to our preclinical studies, CAR-T cells strongly eradicated HIV-1-infected target cells making them a particularly suitable candidate to reach a functional HIV cure. In this clinical trial, we mainly intend to evaluate the safety of CAR-T-Cell therapy on HIV patients whose plasma HIV has been successfully suppressed after antiviral therapy.
  Other Names: HIV-1 specific chimeric antigen receptor T cells

SUMMARY:
To evaluate the safety of autologous CAR-T-cell therapy in individuals lived with HIV-1 infection, CAR T cells are infused after ex vivo expansion and transduction with lentiviral vectors encoding a broadly neutralizing HIV-1 scFv antibody.

DETAILED DESCRIPTION:
This study is a prospective, single-center, single-arm, open-label and phase I clinical trial. Subjects with CD4+T cell counts greater than 350/μl and viral loads of <50 copies/ml over 1 year by antiviral treatment are enrolled. T cells are stimulated with CD3 and CD28, transduced with lentiviral vectors encoding a broadly neutralizing HIV-1 scFv antibody and expanded for approximately 2 weeks. Then, patients are infused with CAR T cells at a dosage of 1×10^5 CAR-T cells/kg body weight. If this dose is well tolerated, dosing will be increased to 5×10^5 CAR T cells/kg body weight. After infusion, adverse events, and HIV-1 latent reservoir size and CAR levels in peripheral blood will be monitored to assess the safety of CAR-T-cell treatment, potential therapeutic efficacy and kinetics of CAR T cells.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years
2. HIV-1 infection by confirmed test;
3. Receiving antiviral treatment ≥ 1 years;
4. Current CD4+ T cell count > 350 cells/μl;
5. HIV-1 RNA levels of < 50 copies/ml for at least a year;
6. Patients who agrees to use two effective methods of contraception to avoid pregnancy during the study period.
7. Patients who sign the informed consent form prior to inclusion in the study.

Exclusion Criteria:

1. Patients with concomitant HAV, HBV, HCV, HDV, HEV, EBV, CMV or syphilis infection;
2. A history of AIDS-related opportunistic infections and tumors within 1 year prior to enrollment;
3. A History of corticosteroids or immunosuppressive drugs for autoimmune diseases by physicians within the last 2 years;
4. Participants with clinically significant laboratory abnormalities as follows:

   * Hemoglobin ≤ 10 gm/dl (female), <11g/dl (male)
   * Absolute neutrophil count ≤ 1×10^9/L
   * Platelet count ≤100×10^9/L
   * Alanine aminotransferase (ALT)≥ 2.5 x ULN
   * Aspartate aminotransferase (AST) ≥ 2.5 x ULN
   * Total bilirubin > 1.5 ULN
   * Serum creatinine >110 μmol/L
   * International normalized ratio (INR) >1.5 or activated partial thromboplastin time (APTT) >45 s
5. Patients with severe psychiatric illness, drugs or alcohol abuse;
6. A woman who is in pregnancy or lactation;
7. A history of central nervous system disease, such as cerebral hemorrhage, dementia, epilepsy and autoimmune diseases;
8. Patients with a non-AIDS-related serious underlying disease;
9. Patients who participate in another clinical study currently which may affect the results of this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation the safety of CAR-T-cell treatment | 3 months
  To assess the adverse events of CAR-T-cell therapy in HIV-1 infected individuals by measuring liver function, blood routine, and cytokine and so on in this clinical trial

SECONDARY OUTCOMES:
Assessment the potential therapeutic efficacy of CAR-T cell therapy | 3 months
  To evaluate the change of HIV-1 latent reservoir in peripheral blood after CAR-T-cell therapy by RT-PCR

OTHER OUTCOMES:
Cellular kinetics of CAR-T cells | 3 months
  To measure the cellular kinetics of CAR-T cells after infusion by RT-PCR and flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, MD, Principal Investigator — Beijing 302 Hospital of China
Locations (1):
- 302 Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walker RE, Bechtel CM, Natarajan V, Baseler M, Hege KM, Metcalf JA, Stevens R, Hazen A, Blaese RM, Chen CC, Leitman SF, Palensky J, Wittes J, Davey RT Jr, Falloon J, Polis MA, Kovacs JA, Broad DF, Levine BL, Roberts MR, Masur H, Lane HC. Long-term in vivo survival of receptor-modified syngeneic T cells in patients with human immunodeficiency virus infection. Blood. 2000 Jul 15;96(2):467-74. PMID 10887107
- [Background] Mitsuyasu RT, Anton PA, Deeks SG, Scadden DT, Connick E, Downs MT, Bakker A, Roberts MR, June CH, Jalali S, Lin AA, Pennathur-Das R, Hege KM. Prolonged survival and tissue trafficking following adoptive transfer of CD4zeta gene-modified autologous CD4(+) and CD8(+) T cells in human immunodeficiency virus-infected subjects. Blood. 2000 Aug 1;96(3):785-93. PMID 10910888
- [Background] Abdel-Mohsen M, Richman D, Siliciano RF, Nussenzweig MC, Howell BJ, Martinez-Picado J, Chomont N, Bar KJ, Yu XG, Lichterfeld M, Alcami J, Hazuda D, Bushman F, Siliciano JD, Betts MR, Spivak AM, Planelles V, Hahn BH, Smith DM, Ho YC, Buzon MJ, Gaebler C, Paiardini M, Li Q, Estes JD, Hope TJ, Kostman J, Mounzer K, Caskey M, Fox L, Frank I, Riley JL, Tebas P, Montaner LJ; BEAT-HIV Delaney Collaboratory to Cure HIV-1 infection. Recommendations for measuring HIV reservoir size in cure-directed clinical trials. Nat Med. 2020 Sep;26(9):1339-1350. doi: 10.1038/s41591-020-1022-1. Epub 2020 Sep 7. PMID 32895573
- [Background] Liu B, Zou F, Lu L, Chen C, He D, Zhang X, Tang X, Liu C, Li L, Zhang H. Chimeric Antigen Receptor T Cells Guided by the Single-Chain Fv of a Broadly Neutralizing Antibody Specifically and Effectively Eradicate Virus Reactivated from Latency in CD4+ T Lymphocytes Isolated from HIV-1-Infected Individuals Receiving Suppressive Combined Antiretroviral Therapy. J Virol. 2016 Oct 14;90(21):9712-9724. doi: 10.1128/JVI.00852-16. Print 2016 Nov 1. PMID 27535056
- [Result] Maldini CR, Claiborne DT, Okawa K, Chen T, Dopkin DL, Shan X, Power KA, Trifonova RT, Krupp K, Phelps M, Vrbanac VD, Tanno S, Bateson T, Leslie GJ, Hoxie JA, Boutwell CL, Riley JL, Allen TM. Dual CD4-based CAR T cells with distinct costimulatory domains mitigate HIV pathogenesis in vivo. Nat Med. 2020 Nov;26(11):1776-1787. doi: 10.1038/s41591-020-1039-5. Epub 2020 Aug 31. PMID 32868878